CLINICAL TRIAL: NCT04106739
Title: Auricular Percutaneous Electrical Neural Field Stimulation in Short-Term Treatment of Alcohol Dependence- Neurohaemodynamic Correlates and Feasibility Study
Brief Title: A Study of New Treatment for Excessive Alcohol Users by Electric Stimulation of Nerves Around Ear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DyAnsys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS010
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol dependence; Peripheral electrical nerve field stimulation (PENFS); Auricular nerve stimulation; Vagus nerve stimulation; relapse prevention
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Randomized (permuted block randomization, fixed), Parallel Group, Placebo Controlled Trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Arm (Active Comparator): Active arm: Auricular Percutaneous Electrical Neural Field Stimulation (PENFS) device will stimulate the outer auditory canal. It will deliver with a pulse width of 500 ms. The stimulation frequency pattern is 1.12Hz(hertz), 2.24Hz,4.56Hz, 9.12Hz, 100Hz then 9.12Hz, 4.56Hz,2.28Hz,1.12Hz. This cycle will keep on continuing. An input voltage will be 4.2V(volt).
  Interventions: Device: Drug Relief V(version) 2.0 Auricular Percutaneous Electrical Neural Field Stimulation (PENFS)
- Sham Arm (Sham Comparator): Sham arm: Auricular Percutaneous Electrical Neural Field Stimulation (PENFS) device will stimulate centre of the left ear lobe to a pulse width of 500 ms at same pattern of stimulation frequency mentioned in active PENFS with an input voltage of 4.2V
  Interventions: Device: Drug Relief V(version) 2.0 Auricular Percutaneous Electrical Neural Field Stimulation (PENFS)

INTERVENTIONS:
Device: Drug Relief V(version) 2.0 Auricular Percutaneous Electrical Neural Field Stimulation (PENFS) — This is a Small electronic circuit board with a minimal number of electronic components in it, which is powered by three zinc-air batteries. Each battery consists of 1.4v of charge. From this charge, the circuit produces a maximum voltage of 3.4V under no load condition.
  The produced Voltage is driven as output by using the three stimulation wires, and the fourth insulated wire acts as a ground. The wires are Bio-compatible and do not have any impact when in contact with the human skin. The wire is attached with a needle to transfer the produced voltage into the nerves of the human ear. The sterilized needle (Titanium) is attached at the end of the wire through a snap fit ring. All the materials used are gone through necessary safety and performance testing including bio-compatibility and sterility testing, wherever necessary.

SUMMARY:
Alcohol Use Disorders (AUD's) are a major health and social problem. Relapse is a rule rather than an exception in alcohol dependence, leading to poor outcomes. Craving are frequently associated with relapse. Keeping in mind the high burden of disease due to AUD, limited efficacy of available treatment modalities it is important to study new treatment modalities. Vagus nerve stimulation (VNS) is a promising neuromodulation technique with robust evidence in epilepsy and treatment-resistant depression. fMRI studies show that transcutaneous VNS (tVNS) replicates most of the biological effects of VNS with an additional advantage of being non-invasive. Percutaneous Electrical Neural Field Stimulation (PENFS) of auricular branch of vagus nerve is a variant of tVNS which has shown promise in the treatment of opioid withdrawal. The efficacy of PENFS has been evaluated in AUDs in only handful of studies.

I propose to employ a double-blind randomized sham-controlled trial where 40 subjects with AUD will be randomized to 2 groups, with 1 group receiving 'Active' auricular PENFS, and another group receiving bilateral 'sham' auricular PENFS.

Assessments will be carried out at baseline and after 15 days of advent of PENFS on tasks to assess craving, along with neurohemodynamic changes on functional Magnetic Resonance Image (fMRI). Follow up of patients will be done till the first relapse or till 3 months after the post evaluation, whichever is earlier.

The investigator's hypotheses are:

1. Active PENFS will lead to significantly greater improvement in subjective craving and drinking-related outcomes as compared to sham PENFS in patients with AUD over the follow-up period of 3 months.
2. Active PENFS will produce a significantly differential Blood Oxygen Level Dependent (BOLD) activation-deactivation pattern of brain regions (greater activation of dorsolateral prefrontal cortex and anterior cingulate cortex and along with deactivation of insular cortex) associated with craving during a cue-induction paradigm as compared to sham PENFS in patients with AUD.
3. Active PENFS will result in a significant differential change in resting-state functional connectivity (fMRI measured) within and between addiction-related neural networks as compared to sham PENFS as evaluated with a resting state fMRI analysis in patients with AUD.

DETAILED DESCRIPTION:
Patients will be recruited into the study after obtaining informed consent. The intervention will be started after completion of detoxification, which will be done with Lorazepam using a front-loading regimen and a drug washout period of 5 half-lives (approx. 3 days) will be given so as not to interfere with the stimulation. Amitriptyline 12.5-25mg will be used as rescue medication for sleep difficulty. All subjects will receive psychosocial interventions related to craving management and relapse prevention as per treatment as usual but will not be prescribed any anti-craving agents during the period of the study.The Drug Relief V 2.0 device will be installed after the detoxification and baseline fMRI scan. After installation, it will automatically provide neurostimulation at regular interval. It will be in situ for the next 15 days. After that, it will be removed temporarily for follow-up fMRI scanning.After completion of scanning a new device will be provided. The current research study will follow standard auricular PENFS procedures with established safety. The battery of the device will last for 15 days. Study subjects will be required to visit NIMHANS (National Institute of mental health and neurosciences) every 15 days to replace the old device for a new one. Till 3 months, all the devices will be provided free of costPatients will be followed up as usual on an outpatient basis, and the recent pattern of alcohol use will be inquired into. The follow-up will be done until the patient has a relapse or a maximum period of three months, whichever is earlier.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Alcohol use disorder (AUD) as per DSM(Diagnostic and Statistical Manual of Mental Disorders)-5 by two psychiatrists working in the department of psychiatry NIMHANS.
2. Male gender.
3. Age not less than 18 years and not more than 50 years.
4. At least, moderately severe AUD as ascertained by a score above 16 in Severity of Alcohol dependence questionnaire (SADQ).
5. Right-handedness as assessed with Edinburgh Handedness Inventory.
6. Informed consent and willingness to come for regular follow-ups (once every two weeks) for three months after recruitment in the study.

Exclusion Criteria:

1. Any diagnosis except alcohol dependence syndrome/ Tobacco dependence syndrome (to apply MINI(Mini International Neuropsychiatric Interview) screen).
2. Contra-indications precluding device use-

   2.1 patient with cardiac implants or similar biomedical implants, 2.2 during pregnancy unless medically advised, 2.3 patient with haemophilia 2.4 skin pathology 2.5 patient with diminished mental capability or physical competence about the handling of the device
3. Left/ mixed handedness
4. Contraindications to MRI

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 1. To restrict number of variables in the study.
  2. Prevalence/Availability of women with AUD is low.
Enrollment: 44 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Craving scores | 90 days
  Change in craving scores measured with Penns Alcohol Craving Scale between baseline and equispaced 6 follow-ups (every 15 days) for 3 months.
  Scale Information:
  1. Scale name: Penn Alcohol Craving Scale. It measures craving for alcohol.
  2. It is a 5-item scale. Each item score range is 0 to 6. So, Scale's total score range is 0 to 30.
  3. Score 0 signifies no craving and score 30 signifies maximum craving.
  4. There is no subscale.

SECONDARY OUTCOMES:
Cue-induced craving resting state fMRI | 14 days
  Change in Cue-induced craving as measured by the VICE protocol 6-minute Visual Image Induced Craving for Ethanol (VICE) paradigm fMRI and resting state fMRI neurohemodynamic changes in the dorsolateral prefrontal cortex, anterior cingulate cortex (ACC) and insular cortex (IC) after 14 days PENFS.
  Time-Points are as follows:
  Time 0 is on the day of recruitment. Time 1 is on Day 14 of recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Diptadhi Mukherjee, MBBS,DM, Principal Investigator — National Institute of Mental Health and Neuro Sciences (NIMHANS)
Locations (1):
- National Institute of Mental Health and Neuro sciences(NIMHANS), Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rehm J, Samokhvalov AV, Shield KD. Global burden of alcoholic liver diseases. J Hepatol. 2013 Jul;59(1):160-8. doi: 10.1016/j.jhep.2013.03.007. Epub 2013 Mar 16. PMID 23511777
- [Background] Soyka M, Muller CA. Pharmacotherapy of alcoholism - an update on approved and off-label medications. Expert Opin Pharmacother. 2017 Aug;18(12):1187-1199. doi: 10.1080/14656566.2017.1349098. Epub 2017 Jul 24. PMID 28658981
- [Background] Maisel NC, Blodgett JC, Wilbourne PL, Humphreys K, Finney JW. Meta-analysis of naltrexone and acamprosate for treating alcohol use disorders: when are these medications most helpful? Addiction. 2013 Feb;108(2):275-93. doi: 10.1111/j.1360-0443.2012.04054.x. Epub 2012 Oct 17. PMID 23075288
- [Background] Foxcroft DR, Coombes L, Wood S, Allen D, Almeida Santimano NM. Motivational interviewing for alcohol misuse in young adults. Cochrane Database Syst Rev. 2014 Aug 21;(8):CD007025. doi: 10.1002/14651858.CD007025.pub2. PMID 25140980
- [Background] Koob GF, Volkow ND. Neurocircuitry of addiction. Neuropsychopharmacology. 2010 Jan;35(1):217-38. doi: 10.1038/npp.2009.110. PMID 19710631
- [Background] Schacht JP, Anton RF, Myrick H. Functional neuroimaging studies of alcohol cue reactivity: a quantitative meta-analysis and systematic review. Addict Biol. 2013 Jan;18(1):121-33. doi: 10.1111/j.1369-1600.2012.00464.x. Epub 2012 May 10. PMID 22574861
- [Background] Sutherland MT, McHugh MJ, Pariyadath V, Stein EA. Resting state functional connectivity in addiction: Lessons learned and a road ahead. Neuroimage. 2012 Oct 1;62(4):2281-95. doi: 10.1016/j.neuroimage.2012.01.117. Epub 2012 Feb 1. PMID 22326834
- [Background] Frangos E, Ellrich J, Komisaruk BR. Non-invasive Access to the Vagus Nerve Central Projections via Electrical Stimulation of the External Ear: fMRI Evidence in Humans. Brain Stimul. 2015 May-Jun;8(3):624-36. doi: 10.1016/j.brs.2014.11.018. Epub 2014 Dec 6. PMID 25573069
- [Background] Wang Z, Fang J, Liu J, Rong P, Jorgenson K, Park J, Lang C, Hong Y, Zhu B, Kong J. Frequency-dependent functional connectivity of the nucleus accumbens during continuous transcutaneous vagus nerve stimulation in major depressive disorder. J Psychiatr Res. 2018 Jul;102:123-131. doi: 10.1016/j.jpsychires.2017.12.018. Epub 2017 Dec 28. PMID 29674268
- [Background] Miranda A, Taca A. Neuromodulation with percutaneous electrical nerve field stimulation is associated with reduction in signs and symptoms of opioid withdrawal: a multisite, retrospective assessment. Am J Drug Alcohol Abuse. 2018;44(1):56-63. doi: 10.1080/00952990.2017.1295459. Epub 2017 Mar 16. PMID 28301217
- [Background] Kraus T, Hosl K, Kiess O, Schanze A, Kornhuber J, Forster C. BOLD fMRI deactivation of limbic and temporal brain structures and mood enhancing effect by transcutaneous vagus nerve stimulation. J Neural Transm (Vienna). 2007;114(11):1485-93. doi: 10.1007/s00702-007-0755-z. Epub 2007 Jun 14. PMID 17564758
- [Background] Davidson R. Assessment of the alcohol dependence syndrome: a review of self-report screening questionnaires. Br J Clin Psychol. 1987 Nov;26(4):243-55. doi: 10.1111/j.2044-8260.1987.tb01358.x. PMID 3322456
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar). Br J Addict. 1989 Nov;84(11):1353-7. doi: 10.1111/j.1360-0443.1989.tb00737.x. PMID 2597811
- [Background] Flannery BA, Volpicelli JR, Pettinati HM. Psychometric properties of the Penn Alcohol Craving Scale. Alcohol Clin Exp Res. 1999 Aug;23(8):1289-95. PMID 10470970
- [Background] Stockwell T, Murphy D, Hodgson R. The severity of alcohol dependence questionnaire: its use, reliability and validity. Br J Addict. 1983 Jun;78(2):145-55. doi: 10.1111/j.1360-0443.1983.tb05502.x. No abstract available. PMID 6135435
- [Background] James KE, Bloch DA, Lee KK, Kraemer HC, Fuller RK. An index for assessing blindness in a multi-centre clinical trial: disulfiram for alcohol cessation--a VA cooperative study. Stat Med. 1996 Jul 15;15(13):1421-34. doi: 10.1002/(SICI)1097-0258(19960715)15:133.0.CO;2-H. PMID 8841652